CLINICAL TRIAL: NCT02819726
Title: A Randomized, Double-blind, Parallel Group, Multicenter Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, and Efficacy of SAIT101 Versus MabThera® Versus Rituxan® in Patients With Rheumatoid Arthritis (RA)
Brief Title: PK, PD, Safety, and Efficacy of SAIT101 Versus MabThera® Versus Rituxan® in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Archigen Biotech Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGB001
Record Dates: First submitted 2016-06-20; First posted 2016-06-30 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis
Keywords: an inadequate response to anti -TNF therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: In Part A, patients are randomized in a 1:1:1 ratio to receive one course (baseline and Week 2) of SAIT101 (n=94) versus Rituxan® (n=94) versus MabThera® (n=94).
  At Week 24, patients are evaluated for the second course (Week 24 and 26) of the infusion.
  In Part B, eligible patients in the SAIT101 arm receive the second course of SAIT101 treatment. Eligible patients in the MabThera® arm receive the second course of MabThera® treatment. Eligible patients in the Rituxan® arm are randomized in a 1:1 ratio to receive SAIT101 or Rituxan® treatment. Patients are followed up for safety until Week 52.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAIT101 (Experimental): In Part A, each patient will receive one course of two 1000 mg SAIT101 infusions: one on Day 1 and the second on Day 15. In Part B, patients with an inadequate response (<50% improvement from Baseline in swollen and tender joint count at Week 24) will be eligible for a further course of two 1000 mg infusions of SAIT101 on Week 24 and Week 26.
  Interventions: Biological: SAIT101
- Rituxan (Active Comparator): In Part A, each patient will receive one course of two 1000 mg Rituxan infusions: one on Day 1 and the second on Day 15. In Part B, patients with an inadequate response (<50% improvement from Baseline in swollen and tender joint count at Week 24) will be randomised in a 1:1 ratio to receive Rituxan or SAIT101 10000 mg infusions on Week 24 and Week 26.
  Interventions: Biological: Rituxan
- MabThera (Active Comparator): In Part A, each patient will receive one course of two 1000 mg MabThera infusions: one on Day 1 and the second on Day 15. In Part B, patients with an inadequate response (<50% improvement from Baseline in swollen and tender joint count at Week 24) will be eligible for a further course of two 1000 mg infusions of MabThera on Week 24 and Week 26.
  Interventions: Biological: MabThera

INTERVENTIONS:
Biological: SAIT101 — 1,000 mg i.v. of SAIT101 on Day 1 and 15. 1,000 mg i.v. of SAIT101 on week 24 and 26 for eligible patients.
  Arms: SAIT101
Biological: MabThera — 1,000 mg i.v. of MabThera® on Day 1 and 15. 1,000 mg i.v. of MabThera® on week 24 and 26 for eligible patients.
  Other Names: Rituximab
  Arms: MabThera
Biological: Rituxan — 1,000 mg i.v. of Rituxan® on Day 1 and 15. 1,000 mg i.v. of Rituxan® on week 24 and 26 for eligible patients.
  Other Names: Rituximab
  Arms: Rituxan

SUMMARY:
A randomised, double blind, parallel group, multicentre study yo compare the pharmacokinetics, pharmacokinetics, safety and efficacy of SAIT101 versus MabThera® versus Rituxan® in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel group, multicenter study to compare the pharmacokinetics (PK), pharmacodynamics (PD), safety, efficacy, tolerability, and immunogenicity of SAIT101 (biosimilar rituximab) versus MabThera® versus Rituxan® in patients with rheumatoid arthritis (RA). This study will take place globally across approximately 75 study centers in order to randomize approximately 282 patients. The study consists of Part A from baseline for PK and efficacy analysis, followed by Part B from Week 24 to 52 for safety follow-up in which collects transition data.

ELIGIBILITY:
Inclusion Criteria:

1. Severe RA defined as:

* Diagnosis of RA according to the revised (1987) American College of Rheumatology (ACR) criteria for the classification of RA for at least 3 months prior to screening visit (see Appendix 3).
* And ≥6 swollen joints and ≥6 tender/painful joints (from the 66/68 joint count system).
* And C-reactive protein (CRP) ≥1.0 mg/dL or an erythrocyte sedimentation rate (ESR) ≥28 mm/hour at Screening.
* And positive rheumatoid factor (RF) (≥20 units/mL) or anti cyclic citrullinase peptide (CCP) antibodies (≥10 units/mL) at Screening.

  2. Patients with severe RA who have had an inadequate response to at least 3 months' treatment (according to the approved treatment and dosage) or intolerance (at Investigator's discretion and/or experience of intolerable AE or toxicity such as infusion related reaction, hypersensitivity, anaphylaxis or severe toxicity) to anti-tumour necrosis factor (TNF) therapy (experience of severe adverse event (AE) or toxicity).

  3. Current treatment for RA on an outpatient basis:
* Receiving methotrexate (MTX) 7.5 - 25mg/week (oral or parenteral) for at least 12 weeks, including the last 4 weeks prior to Day 1 at a stable dose, via the same route of administration, dose, and formulation. Patients receiving a lower dose of MTX (<10 mg/week), stable for 4 weeks prior to Day 1, should be doing so as a result of a documented evidence of intolerance to higher doses of MTX.

Exclusion Criteria:

1. Females who are pregnant, breastfeeding, or planning a pregnancy during the Treatment Period of and 12 months after the last infusion of study drug.
2. Class IV as per the Classification of Global Functional Status in Rheumatoid Arthritis (as per ACR 1991 Revised Criteria) (see Appendix 4) or wheelchair/bed bound.
3. History of or current inflammatory joint disease other than RA (including but not limited to gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy or Lyme disease).
4. History of or current systemic autoimmune disorder (including but not limited to systemic lupus erythematosus, inflammatory bowel disease, pulmonary fibrosis, Felty syndrome, scleroderma, inflammatory myopathy, fibromyalgia, juvenile idiopathic arthritis, mixed connective tissue disease, vasculitis or other overlap syndrome), with the exception of the secondary Sjögren's syndrome.
5. Primary or secondary immunodeficiency (history of, or currently active), including known history of human immunodeficiency virus (HIV) infection or positive test at screening.
6. History of opportunistic infection.
7. History of deep space/tissue infection (e.g., fasciitis, abscess, osteomyelitis) and infected prosthetic joint.
8. Active infection of any kind (excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. anti infective agents within 4 weeks prior to Screening or oral anti-infective agents within 2 weeks prior to Screening or use of antibiotic therapy three or more times in the last six months prior to Screening
9. Positive serological test for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C serology.

   * Patients with a negative HBsAg and positive HBcAb must have a hepatitis B virus (HBV) deoxyribonucleic acid (DNA) level <20 IU/mL (or 112 copies/mL) by polymerase chain reaction (PCR). These HBV patients must be willing to undergo monthly PCR HBV DNA testing during treatment and may participate following consultation with a hepatitis expert regarding monitoring and use of HBV antiviral therapy, and provided they agree to receive treatment as indicated. An HBV re-test will be performed monthly including Day 1, Weeks 4, 8, 12, 16, 20, 24, 36, 52, and unscheduled visit if required.
   * Patients with a positive test because of HBV vaccine may be included (i.e., anti-HBs+ and anti HBc-).
   * Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV ribonucleic acid (RNA).
10. Confirmed current active tuberculosis (TB). • Patients with latent TB as determined by positive QuantiFERON-TB test may be enrolled if such patients have written confirmation from health care provider (e.g., Pulmonologist or Infection Specialist) of adequate prophylaxis before or within the screening period and no evidence of tuberculosis on a chest X-ray performed within 3 months from Day 1.

    • Screening period can be extended to 60 days for prophylaxis of latent TB.

    • QuantiFERON-TB test can be re-tested, if inconclusive.
11. Any significant cardiac disease (e.g., coronary artery disease with unstable angina, coronary heart failure New York Heart Association Class III and IV, familial long QT syndrome, uncontrolled cardiac disease).
12. History of moderate to severe chronic obstructive pulmonary disease (COPD) and/or history of severe COPD exacerbation(s) within the last 12 months of Screening.
13. Vaccination with live or attenuated vaccines within 6 weeks prior to first dose of study drug or planned administration during study participation or within 4 weeks following last dose of study drug. Treatment with IV Gamma Globulin or the Prosorba® Column within 6 months prior to Day 1.
14. History of a severe allergic reaction or anaphylactic reaction to a biological agent or history of hypersensitivity to any component of the study drug including known hypersensitivity or allergy to a murine product.
15. Hypogammaglobulinemia at screening (Immunoglobulin G (IgG) <600 mg/dL).
16. Patients with hemoglobin <8.5 g/dL, absolute neutrophil count (ANC) <1,500 cells/µL or platelet count <75,000 cells/µL at Screening. If a patient has findings marginally below this limit, re testing is allowed, at the Investigator's discretion, within the 30 day period between Visit 1 and Visit 2.

• Creatinine clearance < 50 mL/min (Cockcroft-Gault formula)

• Liver function: Total bilirubin >2.0 mg/dL (>34 µmol/L) except for patients with Gilbert's Syndrome or hemolysis. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >3 × upper limit of normal (ULN). Patients with total bilirubin >2.0 mg/dL possibly due to Gilbert's Syndrome should have a direct bilirubin checked. If the direct bilirubin is normal and medical history is suggestive/positive for Gilbert's Syndrome, the patient successfully meets the criteria.

The AST and ALT may be repeated once within the Screening period if the initial result exceeds this limit, and the lesser value accepted if it meets this criterion.

18. History of cancer within the last 5 years prior to Screening, treated with anti-cancer chemotherapy, including solid tumors and hematologic malignancies and carcinoma in situ (except basal cell and squamous cell carcinomas of the skin or carcinoma in situ of the cervix uteri that have been excised and cured).

19. Major surgical procedure within 4 weeks prior to or planned within 24 weeks of Day 1, with the exception of surgical procedures for dental prosthesis.

20. Previous treatment with a B cell modulating or B cell depletion therapy, such as, but not limited to rituximab, belimumab, atacicept, tabalumab, ocrelizumab, ofatumumab, obinutuzumab, epratuzumab and other experimental treatments.

21. Injectable corticosteroids within 6 weeks prior to Day 1.

22. Participation in a previous clinical study within 4 weeks of Screening or having received treatment with a drug that has not received regulatory approval for any indication within a minimum of 5 half-lives prior to Day 1.

23. Patients who, based on the Investigator's judgment, have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Conditions may also include cardiovascular, vascular, pulmonary, hepatic, renal, endocrine or neurological conditions as determined by medical history, physical examination, laboratory tests or electrocardiogram (ECG).

24. Patients who, in the judgment of the Investigator, are likely to be non-compliant or uncooperative during the study.

25. History of substance abuse (alcohol or drug).

26. History of demyelinating disorders (such as multiple sclerosis or Guillain-Barré syndrome).

27. Patients at risk of progressive multifocal leukoencephalopathy (PML):

* Patients with immune deficiency such as transplant patients on immunosuppressive medications
* Patients receiving certain kinds of chemotherapy
* Patients receiving natalizumab (Tysabri®) for multiple sclerosis
* Patients with psoriasis on longer term efalizumab (Raptiva®) or patients with acquired immunodeficiency syndrome (AIDS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (14):
  - Research Site, Anniston, Alabama
  - Research Site, El Cajon, California
  - Research Site, La Mesa, California
  - Research Site, Lakewood, California
  - Research Site-1, Los Angeles, California
  - Research Site-2, Los Angeles, California
  - Research Site, San Leandro, California
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Boise, Idaho
  - Research Site, Kansas City, Kansas
  - Research Site, Lansing, Michigan
  - Research Site, Waco, Texas
  - Research Site, Tacoma, Washington
- Bosnia and Herzegovina (2):
  - Research Site, Mostar
  - Research site, Sarajevo
- Bulgaria (3):
  - Research Site-1, Plovdiv
  - Research Site-2, Plovdiv
  - Research Site, Sofia
- Czechia (4):
  - Research site, Brno
  - Research site, Ostrava
  - Research site, Prague
  - Research site, Uherské Hradiště
- Germany (6):
  - Research site, Bad Doberan, Mecklegurg-Vorpommern
  - Research site, Ratingen, North Rhine-Westphalia
  - Research site, Dresden, Saxony
  - Research site, Vogelsang, Saxony-Anhalt
  - Research site, Hamburg
  - Research site, Rendsburg
- Research Site, Budapest, Hungary
- India (6):
  - Research site, Bangalore, Karnataka
  - Research site, Hubli, Karnataka
  - Research site, Pune, Maharashtra
  - Research site, Bikaner, Rajasthan
  - Research site, Jaipur, Rajasthan
  - Research site, Kolkata, West Bengal
- Mexico (2):
  - Research Site, Durango
  - Research Site, Mexico City
- Poland (10):
  - Research site, Gdansk
  - Research site, Krakow
  - Research site, Kłodzko
  - Research site, Nowa Sól
  - Research site, Oświęcim
  - Research site, Poznan
  - Research site, Tychy
  - Research site, Warsaw
  - Research site, Wroclaw
  - Research site, Zamość
- South Korea (8):
  - Research Site, Anyang
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Jeju City
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (3):
  - Research Site, A Coruña
  - Research Site, Fuenlabrada
  - Research Site, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a global study conducted in 66 study centres. The first participant entered the study on 11 October 2016 and the date of the last participants last study visit was 07 November 2018.
Groups:
- SAIT101 (Part A and B): 1000 mg intravenous (iv) SAIT101 on Day 1 and 15 (Part A). 1000 mg iv SAIT101 on week 24 and 26 (Part B) for eligible participants,
- MabThera (Part A and B): 1000 mg iv MabThera on Day 1 and 15 (Part A). 1000 mg iv MabThera on week 24 and 26 (Part B) for eligible participants.
- Rituxan (Part A and B): 1000 mg iv of Rituxan on Day 1 and 15 (Part A). 1000 mg iv of Rituxan on week 24 and 26 (Part B) for eligible participants
- SAIT101 (Part B Only): 1000 mg iv SAIT101 on week 24 and 26 (Part B) for eligible participants,
Period: Part A (All Participants)
Arm/Group | SAIT101 (Part A and B) | MabThera (Part A and B) | Rituxan (Part A and B) | SAIT101 (Part B Only)
Started (Received at least 1 infusion of study treatment in Part A) | 98 | 98 | 98 | 0
Completed | 92 | 88 | 87 | 0
Not Completed | 6 | 10 | 11 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 6 | 0
Not completed — Protocol non-compliance | 3 | 4 | 5 | 0
Period: Part B (All Participants)
Arm/Group | SAIT101 (Part A and B) | MabThera (Part A and B) | Rituxan (Part A and B) | SAIT101 (Part B Only)
Started (Received at least 1 infusion of treatment in Part B. 220 participants were re-treated in Part B) | 73 (19 participants who completed Part A were not eligible for Part B) | 70 (18 participants completing Part A were not eligible for Part B) | 39 (5 participants completing Part A were ineligible for Part B.) | 38 (5 participants completing Part A were ineligible for Part B.)
Completed | 70 | 68 | 35 | 36
Not Completed | 3 | 2 | 4 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Not completed — Protocol non-compliance | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SAIT101: SAIT101: 1,000 mg i.v. of SAIT101 on Day 1 and 15. 1,000 mg i.v. of SAIT101 on week 24 and 26 for eligible participants.
- MabThera: MabThera: 1,000 mg i.v. of MabThera® on Day 1 and 15. 1,000 mg i.v. of MabThera® on week 24 and 26 for eligible participants.
- Rituxan: Rituxan: 1,000 mg i.v. of Rituxan® on Day 1 and 15. 1,000 mg i.v. of Rituxan® on week 24 and 26 for eligible participants.
- Total: Total of all reporting groups
Arm/Group | SAIT101 | MabThera | Rituxan | Total
Number analyzed (Participants) | 98 | 98 | 98 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.41) | 52.5 (10.87) | 52.1 (12.09) | 51.8 (11.79)
Age, Customized [Count of Participants; unit: Participants]
  18-60 years | 76 | 75 | 71 | 222
  >60 years | 22 | 23 | 27 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 81 | 80 | 240
  Male | 19 | 17 | 18 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 30 | 29 | 89
  Not Hispanic or Latino | 68 | 68 | 69 | 205
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 20 | 21 | 65
  Asian | 18 | 19 | 24 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 52 | 56 | 52 | 160
  More than one race | 2 | 3 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 5 | 3 | 6 | 14
  Hungary | 3 | 0 | 4 | 7
  Czechia | 7 | 3 | 2 | 12
  United States | 9 | 13 | 6 | 28
  Poland | 15 | 19 | 23 | 57
  Mexico | 27 | 21 | 21 | 69
  Bulgaria | 4 | 5 | 4 | 13
  Bosnia and Herzegovina | 4 | 3 | 1 | 7
  Germany | 2 | 3 | 2 | 8
  India | 13 | 16 | 17 | 46
  Spain | 9 | 12 | 12 | 33
Disease duration [Mean (Standard Deviation); unit: years] | 9.8 (6.73) | 11.2 (7.72) | 9.3 (7.10) | 10.1 (7.22)
C-reactive protein [Mean (Standard Deviation); unit: mg/L] — C-reactive protein (CRP) level (Mg/L). CRP is a marker for inflammation. a normal reading is <3 Mg/L. Higher values indicate disease related inflammation and increased cardiovascular risk.
  CRP levels between 3 Mg/L and 10 Mg/L are mildly elevated. Levels between 10 Mg/L and 100 Mg/L are moderately elevated and CRP levels above 100 Mg/L are severely elevated.
  mg/L | 19.5 (28.99) | 15.3 (20.63) | 16.2 (17.91) | 17.0 (2.99)
Erythrocyte sedimentation rate [Mean (Standard Deviation); unit: mm/hr] — Population: Results were not available for 1 participant in each treatment arm
  mm/hr
    number analyzed (Participants) | 97 | 97 | 97 | 291
    (all) | 51.0 (26.58) | 47.5 (22.87) | 51.5 (23.35) | 50.0 (24.31)
Swollen Joint Count (SJC66) [Mean (Standard Deviation); unit: Joints] — Population: Results were not available for 1 participant in the MabThera treatment arm
  Joints
    number analyzed (Participants) | 98 | 97 | 98 | 293
    (all) | 15.2 (7.97) | 15.2 (7.01) | 13.0 (6.19) | 14.5 (7.14)
Tender Joint Count (TJC68) [Mean (Standard Deviation); unit: Joints] — Population: Results were not available for 1 participant in the MabThera treatment arm
  Joints
    number analyzed (Participants) | 98 | 97 | 98 | 293
    (all) | 21.7 (11.08) | 22.6 (13.66) | 20.0 (10.84) | 21.4 (11.93)
Patient Global Assessments Visual Analogue Scale (VAS) Score [Mean (Standard Deviation); unit: units on a scale] — Patients global assessment of disease activity (assessed on 1 to 100 mm Visual Analog Scale [VAS]). Where 0 = no disease activity and 100 = maximum disease activity. Population: Results were not available for 1 participant in each treatment arm
  units on a scale
    number analyzed (Participants) | 97 | 97 | 97 | 291
    (all) | 68.9 (15.87) | 67.6 (17.53) | 70.8 (17.04) | 69.1 (16.82)
Physician Global Assessment VAS Score [Mean (Standard Deviation); unit: units on a scale] — Physicians global assessment of disease activity (assessed on 1 to 100 mm Visual Analog Scale [VAS]). Where 0 = no disease activity and 100 = maximum disease activity. Population: Results were not available for 1 participant in the SAIT101 treatment arm and 1 participant in the MabThera treatment arm
  units on a scale
    number analyzed (Participants) | 97 | 97 | 98 | 292
    (all) | 71.0 (14.3) | 69.4 (15.9) | 69.8 (14.32) | 70.1 (14.51)
Patient Pain Assessment VAS Score [Mean (Standard Deviation); unit: units on a scale] — Patients assessment of pain (assessed on 1 to 100 mm Visual Analog Scale [VAS]) where 0 = no pain and 100 = severe pain. Population: Results were not available for 1 participant in the Rituxan treatment arm
  units on a scale
    number analyzed (Participants) | 98 | 98 | 97 | 293
    (all) | 67.0 (18.71) | 68.8 (20.02) | 70.7 (19.06) | 68.8 (19.27)
Health Assessment Questionnaire Disability Index (HAQ-DI) Score [Mean (Standard Deviation); unit: Score] — HAQ-DI contains 20 questions split into 8 categories (dressing & grooming, arising, eating, walking, hygiene, reach, grip & activities).
  Scores were: 0 = Without ANY Difficulty; 1 = With SOME Difficulty; 2 = With MUCH Difficulty; 3 = UNABLE to Do. Total scores were calculated as the summed category scores divided by the number of categories.
  Total HAQ-DI scores are presented which range from 0 to 3. Higher scores represent a worse outcome. Scores of 0 to 1 represent mild to moderate difficulty, 1 to 2 moderate disability, and 2 to 3 severe to very severe disability. Population: Results were not available for 1 participant in the Rituxan treatment arm
  Score
    number analyzed (Participants) | 98 | 98 | 97 | 293
    (all) | 1.7 (0.57) | 1.7 (0.64) | 1.6 (0.64) | 1.7 (0.62)
Disease activity score based on a 28-joint count-C-Reactive Protein (DAS-28-CRP( [Mean (Standard Deviation); unit: units on a scale] — Disease Activity Score 28-C-Reactive Protein (DAS28-CRP) consisted of tender joint counts (TJC), swollen joint counts (SJC) & C-reactive protein (CRP) blood levels. Total DAS28-CRPscores are presented and range from 2.0 (minimum) to 10 (maximum). Lower scores represent a better patient outcome. Disease remission is considered achieved if the score is between 0 and <2.6. Low disease activity corresponds to 2.6 to <3.2. Moderate activity is between 3.2 & ≤5.1, while high activity is above 5.1. Population: Results were not available for 1 participant in the MabThera treatment arm
  units on a scale
    number analyzed (Participants) | 98 | 97 | 98 | 293
    (all) | 5.28 (0.890) | 5.29 (0.807) | 5.17 (0833) | 5.25 (0.843)
Disease activity score based on a 28-joint count - Erythrocyte sedimentation Rate (DAS28-ESR) [Mean (Standard Deviation); unit: units on a scale] — Disease Activity Score 28- Erythrocyte Sedimentation Rate (DAS28-ESR) consisted of tender joint counts (TJC), swollen joint counts (SJC) & erythrocyte sedimentation rate (ESR). The formula is: [0.56*SQRT(tender 28 joint count)+0.28*SQRT(swollen 28 joint count)+0.7*ln(ESR)]+0.014*patient global health assessment.
  Total DAS28-ESR scores are presented. Total scores range from 2 (minimum) to 10 (maximum). A lower score represented a better patient outcome. A DAS28-ESR of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
  . Population: Results were not available for 2 participants in each treatment arm
  units on a scale
    number analyzed (Participants) | 96 | 96 | 96 | 288
    (all) | 6.54 (0.844) | 6.53 (0.781) | 6.48 (0.758) | 6.52 (0.793)
Anti-drug Antibody (ADA) Status Positive [Count of Participants; unit: Participants] — Population: Results were not available for 2 participants in the Rituxan arm
  Participants
    number analyzed (Participants) | 98 | 98 | 96 | 292
    (all) | 2 | 1 | 4 | 7
Height [Mean (Standard Deviation); unit: cm] — Population: Results were not available for 1 participant in the Rituxan treatment arm
  cm
    number analyzed (Participants) | 98 | 98 | 97 | 293
    (all) | 162.6 (9.29) | 161.3 (8.79) | 163.3 (8.37) | 162.4 (8.83)
Weight [Mean (Standard Deviation); unit: kg] | 73.0 (17.62) | 71.9 (16.94) | 71.6 (17.99) | 72.2 (17.47)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Population: Results were not available for 1 participant in the Rituxan treatment arm
  Kg/m^2
    number analyzed (Participants) | 98 | 98 | 97 | 293
    (all) | 27.5 (5.48) | 27.5 (5.46) | 26.7 (5.95) | 27.2 (5.63)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Cure From Time 0 to Last Quantifiable Concentration (AUC0-t)
Description: Pharmacokinetic endpoint: Area under the concentration-time curve from time 0 (immediately predose on Day 1) to last quantifiable concentration (AUC0-t). Geometric means by treatment (Pharmacokinetic Analysis Set).
Time Frame: Samples for pharmacokinetic evaluation were taken at Baseline and Weeks 0, 1, 2, 3, 4, 8, 12, 16, 20 and 24. Unscheduled visit samples were taken at the discretion of the investigator.
Population: Pharmacokinetic Analysis Set. (AUC(0-t) could not be determined for 15 participants in the SAIT101 arm, 23 participants in the MabThera arm and 17 in the Rituxan arm as the Week 24 sample was either collected post-dose (i.e. not evaluable), was out of the collection window or was missing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Groups:
- SAIT101: 1000 mg intravenous (iv) SAIT101 on Day 1 and 15 (Part A). 1000 mg iv SAIT101 on week 24 and 26 (Part B) for eligible participants,
- MabThera: 1000 mg iv MabThera on Day 1 and 15 (Part A). 1000 mg iv MabThera on week 24 and 26 (Part B) for eligible participants.
- Rituxan: 1000 mg iv of Rituxan on Day 1 and 15 (Part A). 1000 mg iv of Rituxan on week 24 and 26 (Part B) for eligible participants
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 79 | 70 | 76
h*µg/mL | 144500 (34.2) | 151600 (33.2) | 154600 (35.6)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; The statistical comparison of the loge-transformed primary parameters between treatments is based on an analysis of variance model (ANOVA) with fixed effect for treatment; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ration = 95.33, 90% CI 2-sided [87.07 to 104.37]
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; The statistical comparison of the loge-transformed primary parameters between treatments is based on an analysis of variance (ANOVA) model with fixed effect for treatment; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 93.43, 90% CI 2-sided [85.54 to 102.15]
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 98.06, 90% CI 2-sided [89.49 to 107.45]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC0-∞)
Description: Pharmacokinetic endpoint: Area Under the Plasma Concentration from time 0 to infinity (AUC0-∞ (infinity). Calculated by linear up/log down trapezoidal summation and extrapolated to infinity by addition of the last quantifiable concentration divided by the elimination rate constant: AUC(0-last) + C(last)/λz.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set. AUC0-∞ could not be calculated for 1 participant in the SAIT101 arm, 2 participants in the MabThera arm and 2 participants in the Rituxan arm as either the terminal phase was undetermined, the samples were missing or the Regulatory Scientific Quality (RSQ) was <0.800.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 91 | 91
h*µg/mL | 152300 (34.6) | 161900 (32.2) | 161300 (33.3)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 94.07, 90% CI 2-sided [86.91 to 101.81]
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ration = 94.39, 90% CI 2-sided [87.21 to 102.16]
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 100.35, 90% CI 2-sided [92.68 to 108.65]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC0-D15)
Description: Pharmacokinetic endpoint: Area Under the Concentration verses time from time 0 to Day 15 prior to infusion (AUC0-D15) calculated by linear up/log down trapezoidal summation. Actual time/concentration on Day 15 was used for the calculation of this parameter unless the parameter was derived by interpolation.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set. AUC0-D15 could not be determined for 3 participants in the SAIT101 arm, 5 participants in the MabThera arm and 10 participants in the Rituxan arm as either the 336-hours blood sample was collected <312 hours or samples were missing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 91 | 88 | 83
h*µg/mL | 42950 (26.7) | 44600 (25.6) | 43540 (24.1)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 96.31, 90% CI 2-sided [90.52 to 102.46]
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 98.65, 90% CI 2-sided [92.64 to 105.05]
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 102.43, 90% CI 2-sided [96.14 to 109.14]

4. Primary Outcome: Peak Plasma Concentration (Cmax) After Day 15 Infusion
Description: Pharmacokinetic endpoint: Maximum Plasma Concentration (Cmax) after Day 15 infusion (Dose 2)
Time Frame: Samples for pharmacokinetic evaluation were taken at Baseline and Weeks 0, 1 and 2 (Pre-dose 2). Unscheduled visit samples were taken at the discretion of the investigator.
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 94 | 93 | 93
µg/mL | 406.0 (28.3) | 427.7 (28.3) | 411.1 (24.5)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 94.93, 90% CI 2-sided [89.03 to 101.23]
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 98.75, 90% CI 2-sided [92.61 to 105.30]
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 104.03, 90% CI 2-sided [97.54 to 110.95]

5. Primary Outcome: Trough Concentration (Ctrough) Before the Second Infusion on Day 15
Description: Pharmacokinetic endpoint: Trough concentration (Ctrough) before the second infusion on Day 15 (Dose 2). Trough (pre-dose) concentration prior to second infusion on Day 15 obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 4
Population: Pharmacokinetic Analysis Set. Ctrough could not be determined for 11 participants in the SAIT101 arm, 12 participants in the MabThera arm and 16 participants in the Rituxan arm as samples were collected outside of a 312 to 360 hour window.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 83 | 81 | 77
µg/mL | 60.35 (40.3) | 67.75 (36.2) | 58.84 (97.9)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 89.08, 90% CI 2-sided [77.20 to 102.79]
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 102.56, 90% CI 2-sided [88.72 to 118.56]
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%) for all treatment comparisons; GLS Mean Ratio = 115.13, 90% CI 2-sided [99.51 to 133.21]

6. Primary Outcome: Change From Baseline in DAS28-CRP at Week 24
Description: Disease Activity Score 28 C-reactive protein score (DAS28-CRP) at Week 24 (Full Analysis Set). CRP samples were collected at Baseline and Weeks 8, 16 and 24. DAS28-CRP was calculated using the following equation: [0.56*Square Root (SQRT) (tender 28 joint count)+0.28*SQRT(swollen 28 joint count)+0.36*ln(CRP+1)]*1.10+1.15.
  Total DAS28-CRP scores were calculates and range from 2.0 (minimum) to 10 (maximum). Lower scores represent a better patient outcome. Disease remission is considered achieved if the score is between 0 and <2.6. Low disease activity corresponds to 2.6 to <3.2. Moderate activity is between 3.2 & ≤5.1, while high activity is above 5.1.
Time Frame: Baseline and Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 91 | 87 | 85
Score on a scale | -0.991 (1.1735) | -0.832 (0.8483) | -0.861 (0.9488)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Least square means and confidence intervals (CIs) were estimated from an ANCOVA model containing treatment group as a factor and baseline DAS28-CRP value as a covariate. ANCOVA model contains treatment group only; Test type: Equivalence — The equivalence between 2 study treatments would be declared if the two-sided 95% CI of the difference in change from baseline in DAS28-CRP at week 24 in entirely contained within the equivalence margin of [-0.6,0.6]; p = 0.2402, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.422 to 0.106], Standard Error of Mean 0.134
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; Least square means and CIs were estimated from an ANCOVA model containing treatment group as a factor and baseline DAS28-CRP value as a covariate. ANCOVA model contains treatment group only; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.1346, ANCOVA; LS Means Difference = -0.20, 95% CI 2-sided [-0.469 to 0.063], Standard Error of Mean 0.135
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 6, analysis 2]; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.7429, ANCOVA; LS Means Difference = -0.04, 95% CI 2-sided [-0.314 to 0.224], Standard Error of Mean 0.137

7. Secondary Outcome: Area Under the Concentration Time Curve Week 2 to Week 24 (AUC(w2-24)
Description: Pharmacokinetic endpoint: Area under the concentration time curve week 2 to week 24 (AUC(w2-24) calculated by linear up/log down trapezoidal summation.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set. AUC0-w24 could not be determined for 30 participants in the SAIT101 arm, 32 participants in the MabThera arm and 28 participants either in the Rituxan arm as either there was no concentration at the start and/or end time, the Week 24 sample was out of window or samples were missing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 64 | 61 | 65
h*µg/mL | 107300 (41.1) | 109200 (40.0) | 116000 (40.2)

8. Secondary Outcome: Area Under the Concentration Time Curve Day 0 to Week 12 (AUC(0-w12))
Description: Pharmacokinetic endpoint: Area under the concentration time curve Day 0 to Week 12 calculated by linear up/log down trapezoidal summation.
Time Frame: Samples for pharmacokinetic evaluation were taken at Baseline and Weeks 0, 1, 2, 3, 4, 8 and 12. Unscheduled visit samples were taken at the discretion of the investigator.
Population: Pharmacokinetic Analysis Set. AUC0-w12 could not be determined for 1 participant in the SAIT101 arm, 4 participants in the MabThera arm and 1 participant in the Rituxan arm because samples were missing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 89 | 92
h*µg/mL | 148500 (33.1) | 157400 (30.3) | 155900 (33.1)

9. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) (Dose 1)
Description: Pharmacokinetic endpoint: Maximum plasma concentration over the first dosing interval obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set. Tmax (dose 1) could not be determined for 1 participant in the SAIT101 arm, 1 patient in the MabThera arm and 2 participants in the Rituxan arm as samples were missing or set to missing due to initial or embedded Below the Limit of Quantification (BLQ)..
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 92 | 91
Hours | 5.167 [3.00 to 6.50] | 5.167 [3.00 to 358.75] | 4.500 [3.00 to 6.75]

10. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) (Dose 2)
Description: Time of maximum concentration postinfusion over the second dosing interval, obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 94 | 93 | 93
Hours | 4.167 [2.92 to 5.50] | 4.167 [0.00 to 48.08] | 4.250 [2.92 to 23.50]

11. Secondary Outcome: Apparent Terminal Rate Constant (λz)
Description: Pharmacokinetic endpoint: Apparent terminal rate constant (λz) determined by linear regression of the terminal points of the log-linear concentration-time curve. Best fit method followed by visual assessment was used to identify the terminal linear phase of the concentration-time profile. A minimum of 3 data points was used for determination.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set. λz could not be determined for 1 participant in the SAIT101 arm, 2 participants in the MabThera arm and 1 participant in the Rituxan arm as either the terminal phase was undetermined or the Regulatory Scientific Quality (RSQ) was <0.800.
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 91 | 92
1/hr | 0.002358 (0.00061132) | 0.002283 (0.00067311) | 0.002240 (0.00059435)

12. Secondary Outcome: Systemic Clearance (CL)
Description: Pharmacokinetic endpoint: Systemic clearance (CL) over the first dosing period calculated as dose (first + second dose) divided by AUC(0-∞).
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set. CL could not be determined for 1 participant in the SAIT101 arm, 2 participants in the MabThera arm and 2 participants in the Rituxan arm as either the terminal phase was undetermined or the Regulatory Scientific Quality (RSQ) was <0.800.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 91 | 91
L/day | 0.01314 (34.6) | 0.01235 (29.0) | 0.01240 (33.3)

13. Secondary Outcome: Volume of Distribution (VD)
Description: Pharmacokinetic endpoint: Volume of distribution (VD) over the first dosing period calculated as dose (first + second dose) divided by [λz AUC(0-∞)]
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set. VD could not be determined for 1 participant in the SAIT101 arm, 2 participants in the MabThera arm and 2 participants in the Rituxan arm as either the terminal phase was undetermined or the Regulatory Scientific Quality was <0.800.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres (L)
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 91 | 91
Litres (L) | 5.757 (28.0) | 5.635 (23.6) | 5.727 (22.9)

14. Secondary Outcome: Terminal Half-life (T1/2)
Description: Pharmacokinetic endpoint: Terminal half-life determined as ln2/λz.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set. T1/2 could not be determined for 1 participant in the SAIT101 arm, 2 participants in the MabThera arm and 1 participant in the Rituxan arm as either the terminal was undetermined or the Regulatory Scientific Quality was <0.800.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 91 | 92
Hours | 303.7 (26.1) | 316.1 (29.0) | 319.7 (26.2)

15. Secondary Outcome: Change From Baseline in DAS28-CRP at Weeks 8, 16, 36 and 52
Description: Disease Activity Score 28-C-Reactive Protein (DAS28-CRP) samples taken at Baseline and Weeks 8, 16, 24, 36 and 52. DAS28-CRP was calculated using the following equation: [0.56*Square Root (SQRT) (tender 28 joint count)+0.28*SQRT(swollen 28 joint count)+0.36*ln(CRP+1)]*1.10+1.15.
  Total DAS28-CRP scores are presented and range from 2.0 (minimum) to 10 (maximum). Lower scores represent a better patient outcome. Disease remission is considered achieved if the score is between 0 and <2.6. Low disease activity corresponds to 2.6 to <3.2. Moderate activity is between 3.2 & ≤5.1, while high activity is above 5.1.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: Full Analysis Set (analyses are reported in terms of the arm that the patient was initially randomised into. In the Rituxan arm only, patients eligible for treatment in Part B underwent a second randomisation to receive either Rituxan or SAIT101 and are reported in the Rituxan arm according to their initial randomisation).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 97 | 98
score on a scale
  Day 1 (Baseline) | 5.282 (0.8899) | 5.288 (0.8073) | 5.170 (0.8326)
  Week 8: number analyzed (Participants) | 93 | 93 | 93
  Week 8 | 4.405 (1.0189) | 4.324 (1.1132) | 4.251 (1.1392)
  Week 16: number analyzed (Participants) | 93 | 93 | 92
  Week 16 | 4.001 (1.1116) | 4.155 (0.9750) | 4.100 (1.0044)
  Week 24: number analyzed (Participants) | 91 | 88 | 85
  Week 24 | 4.300 (1.0331) | 4.463 (1.0648) | 4.443 (0.9774)
  Week 36: number analyzed (Participants) | 90 | 83 | 84
  Week 36 | 3.552 (1.1452) | 3.823 (0.9290) | 3.716 (1.0684)
  Week 52 (End of Study(: number analyzed (Participants) | 92 | 88 | 87
  Week 52 (End of Study( | 3.660 (1.2636) | 3.754 (1.3037) | 3.518 (1.1276)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS). Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and Baseline DAS28-CRP value as a covariate. ANCOVA model contains treatment group only; Test type: Other; p = 0.6068, ANCOVA; LS Means Difference = -0.09, 95% CI 2-sided [-0.428 to 0.250], Standard Error of Mean 0.172
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; Week 52 (EOS) Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and Baseline DAS28-CRP value as a covariate. ANCOVA model contains treatment group only; Test type: Other; p = 0.5990, ANCOVA; LS Means Difference = 0.09, 95% CI 2-sided [-0.249 to 0.430], Standard Error of Mean 0.172
Statistical Analysis 3: Comparison: MabThera vs Rituxan; Week 53 (EOS) MabThera vs Rituxan. Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and Baseline DAS28-CRP value as a covariate. ANCOVA model contains treatment group only; Test type: Other; p = 0.3053, ANCOVA; LS Means Difference = 0.18, 95% CI 2-sided [-0.165 to 0.532], Standard Error of Mean 0.175

16. Secondary Outcome: American Collage of Rheumatology 20% Response Criteria (ACR20) Response Rates at Weeks 8, 16, 24, 36 and 52
Description: American Collage of Rheumatology (ACR) 20% response criteria (ACR20) response rates were assessed at Baseline and Weeks 8, 16, 24, 36 and 52.
  An ACR20 response is defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [Health Assessment Questionnaire (HAQ)], visual analogue pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
participants
  ACR20 Week 8: number analyzed (Participants) | 95 | 93 | 92
  ACR20 Week 8 | 39 [31.70 to 51.10] | 33 [26.51 to 45.61] | 44 [37.91 to 57.91]
  ACR20 Week 16: number analyzed (Participants) | 94 | 92 | 91
  ACR20 Week 16 | 50 [43.18 to 62.95] | 54 [48.48 to 68.21] | 53 [47.98 to 67.84]
  ACR20 Week 24: number analyzed (Participants) | 92 | 87 | 86
  ACR20 Week 24 | 36 [28.79 to 49.35] | 31 [26.37 to 46.11] | 34 [29.86 to 50.10]
  ACR20 Week 36: number analyzed (Participants) | 90 | 82 | 83
  ACR20 Week 36 | 63 [59.87 to 78.49] | 47 [46.52 to 67.46] | 58 [58.00 to 78.69]
  ACR20 Week 52 (EOS): number analyzed (Participants) | 94 | 90 | 89
  ACR20 Week 52 (EOS) | 60 [53.75 to 72.82] | 49 [44.18 to 64.34] | 59 [55.98 to 75.26]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS) assessment. The 95% CIs for ACR response rate and difference were derived using the Wilson Score method; Test type: Other; Difference (%) = 9.4, 95% CI 2-sided [-4.74 to 23.03], Standard Error of Mean 7.22
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; Week 52 (EOS) assessment. The 95% CIs for ACR response rate and difference were derived using the Wilson Score method; Test type: Other; Difference (%) = -2.5, 95% CI 2-sided [-15.95 to 11.22], Standard Error of Mean 7.05
Statistical Analysis 3: Comparison: MabThera vs Rituxan; Week 52 (EOS) assessment. The 95% CIs for ACR response rate and difference were derived using the Wilson Score method; Test type: Other; Difference (%) = -11.8, 95% CI 2-sided [-25.47 to 2.45], Standard Error of Mean 7.26

17. Secondary Outcome: American Collage of Rheumatology 50% Response Criteria (ACR50) Response Rates and American Collage of Rheumatology 70% Response Criteria (ACR70) at Weeks 8, 16, 24, 36 and 52
Description: Efficacy endpoint: American Collage of Rheumatology 50% response criteria (ACR50) response rates and American Collage of Rheumatology 70% response criteria (ACR70) at weeks 8, 16, 24, 36 and 52.
  An ACR50 response is defined as both improvement of 50% in the number of tender and number of swollen joints, and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [Health Assessment Questionnaire (HAQ)], visual analogue pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
  An ACR70 response is defined as both improvement of 70% in the number of tender and number of swollen joints, and a 70% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [Health Assessment Questionnaire (HAQ)], visual analogue pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
participants
  ACR50 Week 8: number analyzed (Participants) | 95 | 93 | 93
  ACR50 Week 8 | 13 [8.17 to 22.02] | 11 [6.73 to 19.95] | 14 [9.29 to 23.94]
  ACR70 Week 8: number analyzed (Participants) | 95 | 93 | 92
  ACR70 Week 8 | 2 [0.58 to 7.35] | 2 [0.59 to 7.51] | 2 [0.60 to 7.58]
  ACR50 Week 16: number analyzed (Participants) | 94 | 92 | 91
  ACR50 Week 16 | 17 [11.61 to 27.07] | 16 [11.00 to 26.40] | 14 [9.39 to 24.18]
  ACR70 Week 16: number analyzed (Participants) | 94 | 92 | 91
  ACR70 Week 16 | 9 [5.12 to 17.20] | 4 [1.70 to 10.65] | 5 [2.37 to 12.22]
  ACR50 Week 24: number analyzed (Participants) | 92 | 87 | 86
  ACR50 Week 24 | 15 [10.14 to 25.17] | 8 [4.73 to 17.11] | 5 [2.51 to 12.90]
  ACR70 Week 24: number analyzed (Participants) | 92 | 87 | 86
  ACR70 Week 24 | 8 [4.47 to 16.23] | 2 [0.63 to 8.00] | 3 [1.19 to 9.76]
  ACR50 Week 36: number analyzed (Participants) | 90 | 82 | 83
  ACR50 Week 36 | 37 [31.51 to 51.44] | 19 [15.37 to 33.38] | 25 [21.31 to 40.69]
  ACR70 Week 36: number analyzed (Participants) | 90 | 82 | 83
  ACR70 Week 36 | 19 [13.95 to 30.63] | 6 [3.40 to 15.06] | 12 [8.47 to 23.59]
  ACR50 Week 52 (EOS): number analyzed (Participants) | 94 | 90 | 89
  ACR50 Week 52 (EOS) | 35 [28.14 to 47.33] | 25 [19.58 to 37.80] | 30 [24.74 to 44.02]
  ACR70 Week 52 (EOS): number analyzed (Participants) | 94 | 90 | 89
  ACR70 Week 52 (EOS) | 23 [16.89 to 34.05] | 13 [8.64 to 23.16] | 17 [12.28 to 28.48]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; ACR20 Week 52 (EOS) assessment. The 95% CIs for ACR response rate and difference were derived using the Wilson Score method. The adjusted difference and its 95% confidence intervals are from a logistic regression model containing treatment group as a factor and baseline DAS28-CRP value as a covariate; Test type: Other; Difference (%) = 9.5, 95% CI 2-sided [-4.07 to 22.46], Standard Error of Mean 6.87
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; ACR50 Week 52 (EOS) assessment. The 95% CIs for ACR response rate and difference were derived using the Wilson Score method. The adjusted difference and its 95% confidence intervals are from a logistic regression model containing treatment group as a factor and baseline DAS28-CRP value as a covariate; Test type: Other; Difference (%) = 3.5, 95% CI 2-sided [-10.22 to 17.03], Standard Error of Mean 7.07
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 17, analysis 2]; Test type: Other; Difference (%) = -5.9, 95% CI 2-sided [-19.10 to 7.51], Standard Error of Mean 6.88
Statistical Analysis 4: Comparison: SAIT101 vs MabThera; ACR70 Week 52 (EOS) assessment. The 95% CIs for ACR response rate and difference were derived using the Wilson Score method. The adjusted difference and its 95% confidence intervals are from a logistic regression model containing treatment group as a factor and baseline DAS28-CRP value as a covariate; Test type: Other; Difference (%) = 10.0, 95% CI 2-sided [-1.52 to 21.22], Standard Error of Mean 5.78
Statistical Analysis 5: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 17, analysis 4]; Test type: Other; Difference = 5.4, 95% CI 2-sided [-6.69 to 17.13], Standard Error of Mean 6.08
Statistical Analysis 6: Comparison: MabThera vs Rituxan; [analysis description as in outcome 17, analysis 4]; Test type: Other; Difference (%) = -4.7, 92% CI 2-sided [-15.68 to 6.41], Standard Error of Mean 5.58

18. Secondary Outcome: Individual Components of the ACR Improvement Criteria on Day 1 and at Weeks 8, 16, 24, 36 and 52: Swollen Joint Count (SJC) and Tender Joint Count (TJC) (the 66/68 Joint Count System)
Description: Efficacy endpoint: Individual components of the ACR improvement criteria on Day 1 and at weeks 8, 16, 24, 36 and 52: Swollen Joint Count (SJC) and tender joint count (TJC) (the 66/68 joint count system). SJC and TJC assess the level of skeletal disease involvement. The 66/68 Joint Count evaluates 66 joints for swelling and 68 joints for tenderness.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Least Squares Mean (Standard Deviation); unit: Joints
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
Joints
  Swollen Joint Count Day 1: number analyzed (Participants) | 98 | 97 | 98
  Swollen Joint Count Day 1 | 15.2 (7.97) | 15.2 (15.2) | 13.0 (6.19)
  Swollen Joint Count Week 8: number analyzed (Participants) | 95 | 94 | 93
  Swollen Joint Count Week 8 | 8.6 (7.11) | 8.4 (6.62) | 7.7 (5.92)
  Swollen Joint Count 16: number analyzed (Participants) | 94 | 93 | 92
  Swollen Joint Count 16 | 6.5 (4.86) | 7.8 (7.20) | 7.0 (5.37)
  Swollen Joint Count 24: number analyzed (Participants) | 92 | 88 | 87
  Swollen Joint Count 24 | 8.5 (5.13) | 10.0 (5.85) | 10.0 (6.19)
  Swollen Joint Count 36: number analyzed (Participants) | 90 | 83 | 85
  Swollen Joint Count 36 | 4.8 (6.21) | 5.4 (5.72) | 5.7 (5.49)
  Swollen Joint Count Week 52 (EOS): number analyzed (Participants) | 94 | 91 | 90
  Swollen Joint Count Week 52 (EOS) | 5.2 (6.53) | 6.5 (9.46) | 4.6 (5.04)
  Tender Joint Count Day 1: number analyzed (Participants) | 98 | 97 | 98
  Tender Joint Count Day 1 | 21.7 (11.08) | 22.6 (13.66) | 20.0 (10.84)
  Tender Joint Score Week 8: number analyzed (Participants) | 95 | 94 | 93
  Tender Joint Score Week 8 | 13.9 (9.94) | 14.0 (9.94) | 13.5 (10.69)
  Tender Joint Count Week 16: number analyzed (Participants) | 94 | 93 | 92
  Tender Joint Count Week 16 | 11.1 (10.24) | 12.5 (8.36) | 11.8 (9.09)
  Tender Joint Score Week 24: number analyzed (Participants) | 92 | 88 | 87
  Tender Joint Score Week 24 | 13.6 (9.79) | 15.6 (11.94) | 15.2 (11.62)
  Tender Joint Score Week 36: number analyzed (Participants) | 90 | 83 | 85
  Tender Joint Score Week 36 | 8.3 (9.10) | 10.9 (10.68) | 9.6 (10.81)
  Tender Joint Score Week 52 (EOS): number analyzed (Participants) | 94 | 91 | 90
  Tender Joint Score Week 52 (EOS) | 9.3 (9.34) | 11.9 (15.18) | 9.4 (11.41)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Swollen Joint Count (SJC) Week 52 (EOS) assessment. Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate; Test type: Other; p = 0.1997, ANCOVA; LS Means Difference = -1.28, 95% CI 2-sided [-3.230 to 0.671], Standard Error of Mean 0.991
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 18, analysis 1]; Test type: Other; p = 0.9098, ANCOVA; LS Means Difference = -0.11, 95% CI 2-sided [-2.074 to 1.848], Standard Error of Mean 0.996
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 18, analysis 1]; Test type: Other; p = 0.2480, ANCOVA; LS Means Difference = 1.17, 95% CI 2-sided [-0.817 to 3.150], Standard Error of Mean 1.008
Statistical Analysis 4: Comparison: SAIT101 vs MabThera; Tender Joint Count (TJC) Week 52 (EOS) assessment. Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate; Test type: Other; p = 0.1931, ANCOVA; LS Means Difference = -1.96, 95% CI 2-sided [-4.909 to 0.996], Standard Error of Mean 1.500
Statistical Analysis 5: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 18, analysis 1]; Test type: Other; p = -0.77, ANCOVA; LS Means Difference = -0.77, 95% CI 2-sided [-3.722 to 2.184], Standard Error of Mean 1.500
Statistical Analysis 6: Comparison: MabThera vs Rituxan; [analysis description as in outcome 18, analysis 1]; Test type: Other; p = 0.4352, ANCOVA; LS Means Difference = 1.19, 95% CI 2-sided [-1.805 to 4.180], Standard Error of Mean 1.520

19. Secondary Outcome: Individual Components of the ACR Improvement Criteria on Day 1 and at Weeks 8, 16, 24, 36 and 52: Physicians Global Assessment of Disease Activity (Assessed on 1 to 100 mm Visual Analog Scale [VAS])
Description: Efficacy endpoint: Individual Components of the ACR Improvement Criteria on Day 1 and at Weeks 8, 16, 24, 36 and 52: Physicians global assessment of disease activity (assessed on 1 to 100 mm Visual Analog Scale [VAS]). Where 0 = no disease activity and 100 = maximum disease activity.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
score on a scale
  Disease Activty iDay 1: number analyzed (Participants) | 97 | 97 | 98
  Disease Activty iDay 1 | 71.0 (14.30) | 69.4 (15.00) | 69.8 (14.32)
  Disease Activity Week 8: number analyzed (Participants) | 95 | 93 | 91
  Disease Activity Week 8 | 45.6 (20.75) | 43.2 (23.86) | 44.6 (23.28)
  Disease Activtiy Week 16: number analyzed (Participants) | 93 | 93 | 91
  Disease Activtiy Week 16 | 39.2 (20.94) | 39.0 (20.97) | 42.3 (20.89)
  Disease Activity Week 24: number analyzed (Participants) | 91 | 87 | 87
  Disease Activity Week 24 | 47.9 (22.28) | 47.8 (20.25) | 49.0 (22.45)
  Disease Activtiy Week 36: number analyzed (Participants) | 90 | 83 | 86
  Disease Activtiy Week 36 | 30.3 (21.56) | 36.3 (21.71) | 31.4 (20.69)
  Disease Activity Week 52 (EOS): number analyzed (Participants) | 94 | 91 | 90
  Disease Activity Week 52 (EOS) | 31.1 (21.67) | 35.1 (23.49) | 31.2 (22.95)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS) Physician's Disease Activity Assessment. Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate. Change from Study Day 1 (Baseline); Test type: Other; p = 0.2008, ANCOVA; LS Means Difference = -4.16, 95% CI 2-sided [-10.541 to 2.226], Standard Error of Mean 3.242
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; Week 52 (EOS) Physician's Disease Activity Assessment. Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate. Change from Study Day 1 (Baseline; Test type: Other; p = -0.39, ANOVA; LS Means Difference = -0.39, 95% CI 2-sided [-6.771 to 5.994], Standard Error of Mean 3.242
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 19, analysis 2]; Test type: Other; p = 0.2498, ANCOVA; LS Means Difference = 3.77, 95% CI 2-sided [-2.665 to 10.204], Standard Error of Mean 3.268

20. Secondary Outcome: Individual Components of the ACR Improvement Criteria on Day 1 and at Weeks 8, 16, 24, 36 and 52: Participants Assessment of Pain (Assessed on 1 to 100 mm Visual Analog Scale [VAS])
Description: Participants assessment of pain (assessed on 1 to 100 mm Visual Analog Scale [VAS]). Participants assessment of pain (assessed on 1 to 100 mm Visual Analog Scale [VAS]) where 0 = no pain and 100 = severe pain.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
score on a scale
  Assessment of Pain Day 1: number analyzed (Participants) | 98 | 98 | 97
  Assessment of Pain Day 1 | 67.0 (18.71) | 68.8 (20.02) | 68.8 (19.27)
  Assessment of Pain Week 8: number analyzed (Participants) | 95 | 93 | 92
  Assessment of Pain Week 8 | 48.4 (22.79) | 50.4 (22.40) | 47.9 (23.03)
  Assessment of Pain Week 16: number analyzed (Participants) | 94 | 91 | 92
  Assessment of Pain Week 16 | 42.7 (23.34) | 44.6 (20.91) | 44.4 (22.91)
  Assessment of Pain Week 24: number analyzed (Participants) | 92 | 88 | 86
  Assessment of Pain Week 24 | 49.3 (24.15) | 51.6 (21.44) | 51.8 (23.58)
  Assessment of Pain Week 36: number analyzed (Participants) | 90 | 83 | 84
  Assessment of Pain Week 36 | 36.8 (24.56) | 44.9 (23.78) | 41.6 (23.46)
  Assessment of Pain Week 52 (EOS): number analyzed (Participants) | 94 | 91 | 91
  Assessment of Pain Week 52 (EOS) | 41.2 (24.34) | 43.2 (24.42) | 44.5 (26.10)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS) Participants Pain Assessment. Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate. Change from Study Day 1 (Baseline); Test type: Other; p = 0.7322, ANCOVA; LS Means Difference = -1.23, 95% CI 2-sided [-8.0302 to 5.841], Standard Error of Mean 3.592
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 20, analysis 1]; Test type: Other; p = 0.5418, ANCOVA; LS Means Difference = -2.21, 95% CI 2-sided [-9.347 to 4.920], Standard Error of Mean 3.623
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 20, analysis 1]; Test type: Other; p = 0.7869, ANCOVA; LS Means Difference = -0.98, 95% CI 2-sided [-8.136 to 6.169], Standard Error of Mean 3.633

21. Secondary Outcome: Individual Components of the ACR Improvement Criteria on Day 1 and at Weeks 8, 16, 24, 36 and 52: Participants Global Assessment of Disease Activity (Assessed on 1 to 100 mm VAS)
Description: Efficacy endpoint: Individual Components of the ACR Improvement Criteria on Day 1 and at Weeks 8, 16, 24, 36 and 52: Participants global assessment of disease activity (assessed on 1 to 100 mm visual analogue scale [VAS]). Patients rate how their Rheumatoid Arthritis has affected them, where 0 = very well and 100 = very poor.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
score on a scale
  Disease activity Day 1: number analyzed (Participants) | 97 | 97 | 97
  Disease activity Day 1 | 68.9 (15.87) | 67.6 (17.53) | 70.8 (17.04)
  Disease activity Week 8: number analyzed (Participants) | 95 | 94 | 93
  Disease activity Week 8 | 46.9 (22.57) | 49.1 (22.98) | 48.5 (22.93)
  Disease activity Week 16: number analyzed (Participants) | 94 | 93 | 92
  Disease activity Week 16 | 43.9 (21.47) | 44.4 (21.63) | 44.2 (22.82)
  Disease activity Week 24: number analyzed (Participants) | 92 | 88 | 86
  Disease activity Week 24 | 50.8 (23.16) | 51.1 (20.49) | 52.3 (21.90)
  Disease activity Week 36: number analyzed (Participants) | 90 | 82 | 85
  Disease activity Week 36 | 35.7 (22.63) | 42.7 (22.54) | 42.5 (23.70)
  Disease activity Week 52 (EOS): number analyzed (Participants) | 95 | 91 | 91
  Disease activity Week 52 (EOS) | 41.4 (23.02) | 42.4 (24.10) | 43.1 (23.93)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS) Participants Disease Activity Assessment. Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate. Change from Study Day 1 (Baseline); Test type: Other; p = 0.7097, ANCOVA; LS Means Difference = -1.28, 95% CI 2-sided [-8.062 to 5.496], Standard Error of Mean 3.443
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 21, analysis 1]; Test type: Other; p = 0.6683, ANCOVA; LS Means Difference = -1.48, 95% CI 2-sided [-8.280 to 5.317], Standard Error of Mean 3.453
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 21, analysis 1]; Test type: Other; p = 0.9548, ANCOVA; LS Means Difference = -0.20, 95% CI 2-sided [-7.078 to 6.682], Standard Error of Mean 3.494

22. Secondary Outcome: Individual Components of the ACR Improvement Criteria on Day 1 and at Weeks 8, 16, 24, 36 and 52: Participants Assessment of Disability (Health Assessment Questionnaire-Disability Index [HAQ-DI])
Description: the Health Assessment Questionnaire-Disability Index (HAQ-DI) contains 20 questions split into 8 categories (dressing & grooming, arising, eating, walking, hygiene, reach, grip & activities). Scores were: 0 = Without ANY Difficulty; 1 = With SOME Difficulty; 2 = With MUCH Difficulty; 3 = UNABLE to Do. Total scores were calculated as the summed category scores divided by the number of categories.
  Total HAQ-DI scores are presented which range from 0 to 3. Higher scores represent a worse outcome. Scores of 0 to 1 represent mild to moderate difficulty, 1 to 2 moderate disability, and 2 to 3 severe to very severe disability.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
score on a scale
  HAQ-DI Day 1: number analyzed (Participants) | 98 | 98 | 97
  HAQ-DI Day 1 | 1.610 (0.5728) | 1.605 (0.6567) | 1.585 (0.6421)
  HAQ-DI Week 8: number analyzed (Participants) | 95 | 94 | 93
  HAQ-DI Week 8 | 1.168 (0.6318) | 1.314 (0.6919) | 1.176 (0.6398)
  HAQ-DI Week 16: number analyzed (Participants) | 94 | 93 | 92
  HAQ-DI Week 16 | 1.129 (0.5775) | 1.246 (0.6394) | 1.152 (0.6668)
  HAQ-DI Week 24: number analyzed (Participants) | 92 | 88 | 86
  HAQ-DI Week 24 | 1.209 (0.6071) | 1.335 (0.6381) | 1.294 (0.6594)
  HAQ-DI Week 36: number analyzed (Participants) | 90 | 83 | 84
  HAQ-DI Week 36 | 0.994 (0.6220) | 1.182 (0.6883) | 1.061 (0.6247)
  HAQ-DI Week 52 (EOS): number analyzed (Participants) | 94 | 91 | 91
  HAQ-DI Week 52 (EOS) | 1.027 (0.6208) | 1.207 (0.7025) | 1.190 (0.7116)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS) HAQ-DI (0-3). Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate. Change from Study Day 1 (Baseline); Test type: Other; p = 0.0505, ANCOVA; LS Means Difference = -0.14, 95% CI 2-sided [-0.339 to 0.000], Standard Error of Mean 0.086
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 22, analysis 1]; Test type: Other; p = 0.1141, ANCOVA; LS Means Difference = -0.14, 95% CI 2-sided [-0.307 to 0.033], Standard Error of Mean 0.086
Statistical Analysis 3: Comparison: MabThera vs Rituxan; Week 52 (EOS) HAQ-DI )0-3). Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate. Change from Study Day 1 (Baseline); Test type: Other; p = 0.7111, ANCOVA; LS Means Difference = 0.03, 95% CI 2-sided [-0.139 to 0.204], Standard Error of Mean 0.087

23. Secondary Outcome: Individual Components of the ACR Improvement Criteria on Day 1 and at Weeks 8, 16, 24, 36 and 52: C-reactive Protein (CRP) Level
Description: C-reactive protein (CRP) level (Mg/L). CRP is a marker for inflammation. a normal reading is <3 Mg/L. Higher values indicate disease related inflammation and increased cardiovascular risk.
  CRP levels between 3 Mg/L and 10 Mg/L are mildly elevated. Levels between 10 Mg/L and 100 Mg/L are moderately elevated and CRP levels above 100 Mg/L are severely elevated.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Least Squares Mean (Standard Deviation); unit: Mg/L
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
Mg/L
  CRP Day 1 | 19.5 (28.99) | 15.3 (20.63) | 16.2 (17.91)
  CRP Week 8: number analyzed (Participants) | 93 | 93 | 93
  CRP Week 8 | 12.5 (15.78) | 12.3 (20.29) | 10.4 (12.78)
  CRP Week 16: number analyzed (Participants) | 93 | 93 | 92
  CRP Week 16 | 8.5 (11.78) | 7.2 (9.02) | 7.3 (6.90)
  CRP Week 24: number analyzed (Participants) | 91 | 88 | 85
  CRP Week 24 | 9.5 (14.54) | 8.3 (14.40) | 7.9 (10.35)
  CRP Week 36: number analyzed (Participants) | 90 | 83 | 85
  CRP Week 36 | 8.0 (20.33) | 7.0 (10.38) | 7.1 (9.72)
  CRP Week 52 (EOS): number analyzed (Participants) | 92 | 88 | 88
  CRP Week 52 (EOS) | 9.8 (14.14) | 9.1 (14.93) | 7.4 (11.34)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS) CRP. Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline value as a covariate. Change from Study Day 1 (Baseline); Test type: Other; p = 0.8183, ANCOVA; LS Means Difference = -0.43, 95% CI 2-sided [-4.113 to 3.253], Standard Error of Mean 1.871
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 23, analysis 1]; Test type: Other; p = 0.4186, ANCOVA; LS Means Difference = 1.51, 95% CI 2-sided [-2.164 to 5.191], Standard Error of Mean 1.868
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 23, analysis 1]; Test type: Other; p = 0.3035, ANCOVA; LS Means Difference = 1.94, 95% CI 2-sided [-1.768 to 5.655], Standard Error of Mean 1.885

24. Secondary Outcome: Change From Baseline DAS28-erythrocyte Sedimentation Rate (ESR) at Weeks 8, 16, 24, 36 and 52
Description: Disease Activity Score 28- Erythrocyte Sedimentation Rate (DAS28-ESR) consisted of tender joint counts (TJC), swollen joint counts (SJC) & erythrocyte sedimentation rate (ESR). The formula is: [0.56*SQRT(tender 28 joint count)+0.28*SQRT(swollen 28 joint count)+0.7*ln(ESR)]+0.014*patient global health assessment.
  Total DAS28-ESR scores are presented. Total scores range from 2 (minimum) to 10 (maximum). A lower score represents a better patient outcome. A DAS28-ESR of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
score on a scale
  DAS28-ESR Day 1: number analyzed (Participants) | 96 | 96 | 96
  DAS28-ESR Day 1 | 6.537 (0.8440) | 6.533 (.07810) | 6.480 (0.7577)
  DAS28-ESR Week 8: number analyzed (Participants) | 94 | 92 | 93
  DAS28-ESR Week 8 | 5.330 (1.0649) | 5.315 (1.2478) | 5.235 (1.2578)
  DAS28-ESR Week 16: number analyzed (Participants) | 94 | 92 | 92
  DAS28-ESR Week 16 | 4.861 (1.1876) | 5.059 (1.1682) | 4.957 (1.1802)
  DAS28-ESR Week 24: number analyzed (Participants) | 92 | 87 | 85
  DAS28-ESR Week 24 | 5.216 (1.2510) | 5.410 (1.2344) | 5.432 (1.1891)
  DAS28-ESR Week 36: number analyzed (Participants) | 90 | 80 | 80
  DAS28-ESR Week 36 | 4.319 (1.2798) | 4.689 (1.0077) | 4.499 (1.1980)
  DAS28-ESR Week 52 (EOS): number analyzed (Participants) | 92 | 86 | 82
  DAS28-ESR Week 52 (EOS) | 4.435 (1.4375) | 4.485 (1.4390) | 4.391 (1.3947)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 ( EOS) Least square means and confidence intervals were estimated from an ANCOVA model containing treatment group as a factor and baseline DAS28-ESR value as a covariate. ANCOVA model contains treatment group only; Test type: Other; p = 0.9249, ANCOVA; LS Means Difference = 0.02, 95% CI 2-sided [-0.375 to 0.413], Standard Error of Mean 0.200
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 24, analysis 1]; Test type: Other; p = 0.05, ANCOVA; LS Measn Difference = 0.05, 95% CI 2-sided [-0.351 to 0.442], Standard Error of Mean 0.201
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 24, analysis 1]; Test type: Other; p = 0.8962, ANCOVA; LS Means Diference = 0.03, 95% CI 2-sided [-0.376 to 0.430], Standard Error of Mean 0.205

25. Secondary Outcome: Number of Participants With a Major Clinical Response (Continuous ACR70) for at Least 24 Weeks
Description: Efficacy endpoint: number of participants with a major clinical response defined as a continuous ACR70 from Baseline (Day 1) for at least 24 weeks.
  ACR70 is a measure based on American College of Rheumatology criteria of at least a 70% improvement in the number of tender and swollen joints, and a 70% improvement in at least 3 of the following: the patient's global assessment of disease status; the patient's assessment of pain; the patient's assessment of function measured using the Stanford Health Assessment Questionnaire the physician's global assessment of disease status; serum C-reactive protein levels.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
participants
  Major Clinical Response Week 24: number analyzed (Participants) | 92 | 86 | 85
  Major Clinical Response Week 24 | 1 [0.19 to 5.90] | 0 [0.00 to 4.28] | 0 [0.00 to 4.32]
  Major Clinical Response Week 52 (EOS): number analyzed (Participants) | 89 | 81 | 80
  Major Clinical Response Week 52 (EOS) | 2 [0.62 to 7.83] | 0 [0.00 to 4.53] | 1 [0.22 to 6.75]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS) Major Clinical Response. The 95% CIs for major clinical response rate and treatment difference were derived using the Wilson Score method. The adjusted difference and its 95% CI are from a logistic regression model containing treatment group as a factor and baseline DAS28-CRP as a covariate; Test type: Other; Difference (%) = 2.2, 95% CI 2-sided [-2.56 to 7.83], Standard Error of Mean 1.57
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 25, analysis 1]; Test type: Other; Difference (%) = 1.0, 95% CI 2-sided [-4.74 to 6.67], Standard Error of Mean 2.0
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 25, analysis 1]; Test type: Other; Difference (%) = -1.3, 95% CI 2-sided [-6.75 to 3.39], Standard Error of Mean 1.24

26. Secondary Outcome: Number of Participants With a Clinical Remission Response (CRR) at Weeks 8, 16, 24, 36 and 52
Description: Number if Participants with a Clinical Remission Response (CRR) defined by the Simplified Disease Activity Index (SDAI) <3.3 at weeks 8, 16, 24, 36 and 52 (EOS).
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
participants
  CRR Week 8: number analyzed (Participants) | 93 | 92 | 91
  CRR Week 8 | 0 [0.00 to 3.97] | 0 [0.00 to 4.01] | 0 [0.00 to 4.05]
  CRR Week 16: number analyzed (Participants) | 92 | 93 | 91
  CRR Week 16 | 0 [0.00 to 4.01] | 1 [0.19 to 5.84] | 0 [0.00 to 4.05]
  CRR Week 24: number analyzed (Participants) | 90 | 87 | 84
  CRR Week 24 | 0 [0.00 to 4.09] | 1 [0.20 to 6.23] | 0 [0.00 to 4.37]
  CRR Week 36: number analyzed (Participants) | 90 | 82 | 83
  CRR Week 36 | 2 [0.61 to 7.74] | 0 [0.00 to 4.48] | 1 [0.21 to 6.51]
  CRR Week 52 (EOS): number analyzed (Participants) | 92 | 88 | 86
  CRR Week 52 (EOS) | 1 [0.19 to 5.90] | 2 [0.63 to 7.91] | 2 [0.64 to 8.09]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 (EOS). Clinical remission is defined as score of Simplified Disease Activity Index (SDAI) smaller than 3.3. The 95% CIs for clinical remission rate and treatment difference were derived using the Wilson Score method. The adjusted difference and its 95% CI are from a logistic regression model containing treatment group as a factor and baseline DAS28-CRP as a covariate; Test type: Other; Difference (%) = -1.2, 95% CI 2-sided [-6.9 to 3.90], Standard Error of Mean 1.92
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 26, analysis 1]; Test type: Other; Difference (%) = -1.2, 95% CI 2-sided [-7.07 to 3.86], Standard Error of Mean 1.95
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 26, analysis 1]; Test type: Other; Differnce (%) = -0.1, 95% CI 2-sided [-6.05 to 5.83], Standard Error of Mean 2.27

27. Secondary Outcome: Proportion of Participants With European League Against Rheumatism (EULAR) Response at Weeks 8, 16, 24 36 and 52
Description: Efficacy endpoint: Proportion of participants with European League Against Rheumatism (EULAR) response (defined as good response, moderate response or no response) at weeks 8, 16, 24 36 and 52 (EOS). EULAR (European League Against Rheumatism) response was classified using the individual amount of change in the DAS28-CRP score. The DAS28-CRP was classified into 3 categories: low disease activity (<= 3.2), moderate disease activity (> 3.2 and <= 5.1) and high disease activity (> 5.1). Good response was defined as >1.2 improvement in the DAS28-CRP from baseline with low disease activity.
Time Frame: Baseline and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 98 | 98 | 98
participants
  Week 8 Good: number analyzed (Participants) | 93 | 92 | 93
  Week 8 Good | 12 [7.54 to 21.21] | 14 [9.29 to 23.94] | 12 [7.54 to 21.21]
  Week 8 Good or Moderate: number analyzed (Participants) | 93 | 92 | 93
  Week 8 Good or Moderate | 30 [23.62 to 42.30] | 33 [26.82 to 46.05] | 33 [26.51 to 45.61]
  Week 16 Good: number analyzed (Participants) | 93 | 92 | 92
  Week 16 Good | 20 [14.38 to 30.90] | 12 [7.62 to 21.43] | 13 [8.45 to 22.69]
  Week 16 Good or Moderate: number analyzed (Participants) | 93 | 92 | 92
  Week 16 Good or Moderate | 44 [37.47 to 57.36] | 42 [35.85 to 55.80] | 33 [26.82 to 46.05]
  Week 24 Good: number analyzed (Participants) | 91 | 87 | 85
  Week 24 Good | 12 [7.71 to 21.65] | 7 [3.95 to 15.69] | 7 [4.05 to 16.04]
  Week 24 Good or Moderate: number analyzed (Participants) | 91 | 87 | 85
  Week 24 Good or Moderate | 30 [24.17 to 43.14] | 26 [21.28 to 40.19] | 23 [18.76 to 37.34]
  Week 36 Good: number analyzed (Participants) | 90 | 82 | 84
  Week 36 Good | 27 [21.51 to 40.13] | 15 [11.41 to 28.01] | 27 [23.13 to 42.72]
  Week 36 Good or Moderate: number analyzed (Participants) | 90 | 82 | 84
  Week 36 Good or Moderate | 58 [54.15 to 73.56] | 50 [50.00 to 70.82] | 54 [53.62 to 73.70]
  Week 52 (EOS) Good: number analyzed (Participants) | 92 | 87 | 87
  Week 52 (EOS) Good | 34 [27.80 to 47.16] | 31 [26.37 to 46.11] | 32 [27.41 to 47.27]
  Week 52 (EOS) Good or Moderate: number analyzed (Participants) | 92 | 50 | 87
  Week 52 (EOS) Good or Moderate | 59 [53.95 to 73.18] | 50 [46.98 to 67.33] | 63 [62.23 to 80.71]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Week 52 EULAR score 'Good'. EULAR (European League Against Rheumatism) response was classified using the individual amount of change in the DAS28-CRP score. The 95% CIs for EULAR response rate and treatment difference were derived using the Wilson Score method; Test type: Other; Difference (%) = 1.3, 95% CI 2-sided [-12.59 to 15.10], Standard Error of Mean 7.19
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 27, analysis 1]; Test type: Other; Difference (%); Difference (%) = 0.2, 95% CI 2-sided [-13.75 to 14.03], Standard Error of Mean 7.21
Statistical Analysis 3: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 27, analysis 1]; Test type: Other; Difference (%) = -1.1, 95% CI 2-sided [-15.14 to 12.91], Standard Error of Mean 7.29

28. Secondary Outcome: Pharmacodynamic Endpoint: Change From Baseline in Immunoglobulin (IgG, IgM and IgA Levels)
Description: Change from baseline (Day 1) in immunoglobulin G (IgG), Immunoglobulin M (IgM) and Immunoglobulin A (IgA) levels (mg/dL) at Week 8, 16, 24 36 and 52 (End of study)
Time Frame: Baseline (Day 1) and Weeks 8, 16, 24, 36 and 52 (EOS)
Population: Pharmacodynamic Analysis Set (analyses are reported in terms of the arm that the patient was initially randomised into. In the Rituxan arm only, patients eligible for treatment in Part B underwent a second randomisation to receive either Rituxan or SAIT101 and are reported in the Rituxan arm according to their initial randomisation).
Measure: Mean (Standard Deviation); unit: Mg/dL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 95 | 96 | 93
Mg/dL
  IgG Screening | 1231.0 (299.36) | 1230.1 (365.54) | 1203.4 (373.29)
  IgG Week 8: number analyzed (Participants) | 94 | 94 | 91
  IgG Week 8 | 1108.0 (242.20) | 1080.6 (279.75) | 1038.5 (290.01)
  IgG Week 16: number analyzed (Participants) | 91 | 93 | 91
  IgG Week 16 | 1105.2 (232.51) | 1075.7 (277.51) | 1038.5 (290.01)
  IgG Week 24: number analyzed (Participants) | 91 | 83 | 86
  IgG Week 24 | 1114.6 (251.78) | 1077.2 (265.55) | 1023.2 (278.70)
  IgG Week 36: number analyzed (Participants) | 89 | 86 | 84
  IgG Week 36 | 1076.6 (246.62) | 1060.9 (305.12) | 976.6 (249.11)
  IgG Week 52 (EOS): number analyzed (Participants) | 89 | 86 | 87
  IgG Week 52 (EOS) | 1102.0 (274.44) | 1081.1 (285.13) | 999.9 (232.03)
  IgM Screening | 164.3 (76.07) | 167.9 (100.16) | 159.0 (81.36)
  IgM Week 8: number analyzed (Participants) | 94 | 94 | 91
  IgM Week 8 | 137.5 (71.38) | 132.6 (83.58) | 128.9 (68.50)
  IgM Week 16: number analyzed (Participants) | 91 | 94 | 91
  IgM Week 16 | 123.7 (61.08) | 124.9 (85.71) | 117.0 (60.44)
  IgM Week 24: number analyzed (Participants) | 91 | 86 | 86
  IgM Week 24 | 123.3 (62.37) | 117.1 (80.96) | 109.9 (73.11)
  IgM Week 36: number analyzed (Participants) | 89 | 83 | 84
  IgM Week 36 | 111.7 (56.89) | 108.0 (77.79) | 99.7 (56.38)
  IgM Week 52 (EOS): number analyzed (Participants) | 89 | 86 | 87
  IgM Week 52 (EOS) | 109.6 (56.80) | 107.6 (77.00) | 95.2 (52.57)
  IgA Screening | 321.1 (269.22) | 283.4 (134.80) | 342.9 (153.24)
  IgA Week 8: number analyzed (Participants) | 93 | 94 | 93
  IgA Week 8 | 293.6 (176.04) | 264.4 (121.41) | 316.5 (146.15)
  IgA Week 16: number analyzed (Participants) | 91 | 93 | 91
  IgA Week 16 | 301.8 (204.14) | 253.0 (111.58) | 312.7 (151.87)
  IgA Week 24: number analyzed (Participants) | 91 | 86 | 91
  IgA Week 24 | 279.8 (119.87) | 263.0 (121.15) | 307.7 (147.92)
  IgA Week 36: number analyzed (Participants) | 89 | 83 | 89
  IgA Week 36 | 283.8 (204.12) | 259.2 (116.55) | 297.1 (146.85)
  IgA Week 52: number analyzed (Participants) | 89 | 83 | 89
  IgA Week 52 | 269.4 (116.74) | 254.7 (115.38) | 297.8 (138.63)

29. Other Pre Specified Outcome: Pharmacodynamic Endpoint: Depletion of B-lymphocyte Antigen CD19 (CD19+) B-cell Count up to Week 24
Description: Pharmacodynamic endpoint: proportion of participants (n) with depletion of CD19+ B-cell count up to week 24 (Pharmacodynamic analysis set).
Time Frame: Samples for pharmacodynamic evaluation (CD19+ B-cell) were taken at Baseline and Weeks 0, 1, 2, 3, 4, 8, 12, 16, 20 and 24. Unscheduled visit samples were taken at the discretion of the investigator.
Population: Pharmacokinetic data set
Measure: Number; unit: participants
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 95 | 96 | 94
participants | 45 | 46 | 50

30. Other Pre Specified Outcome: Pharmacodynamic Endpoint: Time Needed to CD19+ B-cell Depletion
Description: Time needed to CD19+ B-cell depletion in Part A (calculated as the first time CD19+ B-cell count below 20/µL minus time of first dosing in days).
Time Frame: Samples for pharmacodynamic evaluation (CD19+ B-cell) were taken at Baseline and Weeks 0, 1, 2, 3, 4, 8, 12, 16, 20, 24, 36 and 52. Unscheduled visit samples were taken at the discretion of the investigator.
Population: Pharmacodynamic Analysis Set. Two participants in the SAIT101 arm, 3 participants in the MabThera arm and 3 participants in the Rituxan arm were excluded from the analysis either as they had a depleted C-cell count at baseline and / or if the Week 24 assessment was missing.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 93 | 90
Days | 1.524 (2.6274) | 2.847 (9.1286) | 2.223 (9.0833)

31. Other Pre Specified Outcome: Pharmacodynamic Endpoint: Duration of CD19+ B-cell Depletion
Description: Duration of CD19+ B-cell depletion (only participants that returned to non-depletion at or before week 24 were included)
Time Frame: as for outcome 30
Population: Pharmacodynamic Analysis Set.Pharmacodynamic Analysis Set. Fifty seven participants in the SAIT101 arm, 70 participants in the MabThera arm and 72 participants in the Rituxan arm were excluded from the analysis either as they had a depleted C-cell count at baseline or if the Week 24 assessment was missing.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 36 | 26 | 21
Days | 78.444 (77.5290) | 85.856 (73.4460) | 77.290 (72.0557)

32. Other Pre Specified Outcome: Pharmacodynamic Endpoint: Number of Participants With CD19+ B-cell Count Recover Versus Baseline
Description: Number of participants with CD19+ B-cell count recover versus baseline. Incidence of B-Cell recovery was defined as either CD19+ B-cell counts retuned to baseline or the lower limit or normal of 110 cells/µL at week 24).
Time Frame: as for outcome 30
Population: Pharmacodynamic Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 93 | 93 | 90
Participants | 5 | 4 | 3

33. Other Pre Specified Outcome: Pharmaco Endpoint: Area Under the Concentration Time Curve of CD19 B-cell Count Change at Day 15 and Week 24
Description: Area under the concentration time curve of CD19 B-cell count change at Day 15 (AUEC0-d15) and week 24 (AUEC0-w24) based on change from baseline and percent of baseline values
Time Frame: as for outcome 30
Population: Pharmacodynamic Analysis Set. AUC0-d15 could not be determined for 23 participants in the SAIT101 arm, 20 participants in the MabThera arm and 20 participants in the Rituxan arm as either the baseline data was missing and /or there was a missing b-cell could at the last timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: cells*day/µL)
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 72 | 76 | 73
cells*day/µL)
  AUEC(0-d15) | -2650.0 [-2786.0 to -2513.9] | -2672.1 [-2804.9 to -2539.3] | -2719.4 [-2855.3 to 2583.6]
  AUEC(0-w24): number analyzed (Participants) | 56 | 56 | 52
  AUEC(0-w24) | -32707.6 [-33128.1 to -32287.1] | -33018.3 [-33440.4 to -32596.2] | -33003.7 [-33442.8 to -32564.6]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; The statistical comparison of the between treatments is based on an analysis of covariance (ANOVA) model with fixed effect for treatment and a covariate for baseline value; Test type: Other — Statistical comparison of CD19+ B-cell pharmacokinetic parameters at Day 15 [AUEC(0-d15)]; Statistical Comparisons Difference = 22.1, 90% CI 2-sided [-137.1 to 181.3]
Statistical Analysis 2: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 33, analysis 1]; Test type: Other — Statistical comparison of CD19+ B-cell pharmacokinetic parameters at Day 15 [AUEC(0-d15)]; Statistical Comparisons Difference = 69.5, 90% CI 2-sided [-91.8 to 230.8]
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 33, analysis 1]; Test type: Other — Statistical comparison of CD19+ B-cell pharmacokinetic parameters at Day 15 [AUEC(0-d15)]; Statistical Comparisons Difference = 47.4, 90% CI 2-sided [-112.5 to 207.2]
Statistical Analysis 4: Comparison: SAIT101 vs MabThera; [analysis description as in outcome 33, analysis 1]; Test type: Other — Statistical comparison of CD19+ B-cell pharmacokinetic parameters at Day week [AUEC(0-w24)]; Statistical Comparisons Difference = 310.7, 90% CI 2-sided [-187.9 to 809.4]
Statistical Analysis 5: Comparison: SAIT101 vs Rituxan; [analysis description as in outcome 33, analysis 1]; Test type: Other — Statistical comparison of CD19+ B-cell pharmacokinetic parameters at Day week [AUEC(0-w24)]; Statistical Comparisons Difference = 296.1, 90% CI 2-sided [-213.8 to 806.1]
Statistical Analysis 6: Comparison: MabThera vs Rituxan; [analysis description as in outcome 33, analysis 1]; Test type: Other — Statistical comparison of CD19+ B-cell pharmacokinetic parameters at Day week [AUEC(0-w24)]; Statistical Comparisons Difference = -14.6, 90% CI 2-sided [-527.4 to 498.2]

34. Other Pre Specified Outcome: Pharmacodynamic Endpoint: Change From Baseline in CD19+ B-cell Count During the Study Period
Description: Pharmacodynamic endpoint: Descriptive statistics (mean [SD]) of the change from baseline in CD19+ B-cell count during the study period (Day 15 [AUEC(0-d15] and Week 24 [AUEC(0-w24])
Time Frame: as for outcome 29
Population: Pharmacodynamic Analysis Set. participants in the SAIT101 arm, Twenty three participants in the MabThera arm, 20 participants in the MabThera and 20 participants in the Rituxan arm were excluded from the analysis either as they had a depleted C-cell count at baseline and / or the Week 24 assessment was missing.
Measure: Mean (Standard Deviation); unit: Cells*day/µL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 72 | 76 | 73
Cells*day/µL
  AUEC(0-d15) | -2729 (1915.3) | -2935 (2222.1) | -2367 (1978.1)
  AUEC(0-w24): number analyzed (Participants) | 56 | 56 | 52
  AUEC(0-w24) | -33500 (23881) | -36410 (22883) | -28500 (20878)

35. Other Pre Specified Outcome: Pharmacodynamic Endpoint: Change From Baseline in C-reactive Protein (CRP) Levels at Weeks 8, 16, 24, 36 and 52
Description: Pharmacodynamic endpoint: Change from baseline (Day 1) in C-reactive protein (CRP) levels (mg/dL) at weeks 8, 16, 24, 36 and 52 (EOS)
Time Frame: Baseline (Day 1) and Weeks 8, 16, 24, 26 & 52 (EOS)
Population: Pharmacodynamic Analysis Set
Measure: Mean (Standard Deviation); unit: Mg/dL
Arm/Group | SAIT101 | MabThera | Rituxan
Number analyzed (Participants) | 95 | 96 | 93
Mg/dL
  CRP Day 1 | 19.5 (29.50) | 15.5 (20.76) | 16.1 (17.64)
  CRP Week 8 | 12.5 (15.78) | 12.3 (20.29) | 10.4 (12.85)
  CRP Week 16 | 8.5 (11.78) | 7.2 (9.02) | 7.3 (6.90)
  CRP Week 24 | 9.5 (14.54) | 8.3 (14.40) | 7.9 (10.35)
  CRP Week 36 | 8.0 (10.33) | 7.0 (10.38) | 7.1 (9.72)
  CRP Week 52 (EOS) | 9.8 (14.28) | 9.1 (15.01) | 7.3 (11.33)

ADVERSE EVENTS:
Time Frame: After the participant signed the Informed Consent Form (ICF), but prior to the initiation of study drug, only Serious Adverse Events (SAEs) caused by a protocol mandated procedure should be reported (e.g. SAEs related to invasive procedures such s biopsies). All adverse events were collected for each patient from the start of the first infusion of study drug on Day 1 until the Week 52 Data-cut off.
Description: Safety Analysis Set (analyses are reported in terms of the arm that the patient was initially randomised into. In the Rituxan arm only, patients eligible for treatment in Part B underwent a second randomisation to receive either Rituxan or SAIT101 and are reported in the Rituxan arm according to their initial randomisation).
Arm/Group | SAIT101 | MabThera | Rituxan
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98 | 1/98
Serious Adverse Events (participants affected / at risk) | 7/98 | 7/98 | 13/98
Other Adverse Events (participants affected / at risk) | 39/98 | 37/98 | 43/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAIT101 (N=98) | MabThera (N=98) | Rituxan (N=98)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Oseoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAIT101 (N=98) | MabThera (N=98) | Rituxan (N=98)
Urinary tract infection (Infections and infestations) | 13 (14) | 4 (6) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 8 (10) | 5 (5)
Nasopharyngitis (Infections and infestations) | 7 (9) | 3 (4) | 7 (7)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (7) | 6 (6) | 6 (7)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 8 (9) | 3 (3)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 7 (8)
Hypertension (Vascular disorders) | 2 (2) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT02819726/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT02819726/SAP_001.pdf